CLINICAL TRIAL: NCT07117851
Title: A Prospective, Single-Arm Clinical Study of Disitamab Vedotin Combined With Bicalutamide in HER2 and AR-Expressing Scrotal Paget's Disease
Brief Title: A Study of Disitamab Vedotin + Bicalutamide in HER2/AR-Positive Scrotal Paget's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Fujian Province Tumor Hospital (Other); Qinghai Province Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Ding-Wei Ye, Director of urology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2507324-6
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Extramammary Paget Disease; Scrotum Disease
MeSH Terms: conditions — Paget Disease, Extramammary | interventions — bicalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug: Disitamab Vedotin combined with Bicalutamide (Experimental)
  Interventions: Drug: Disitamab Vedotin combined with Bicalutamide

INTERVENTIONS:
Drug: Disitamab Vedotin combined with Bicalutamide — Single Group Assignment

SUMMARY:
The goal of this clinical trial is to learn if Disitamab Vedotin combined with Bicalutamide works to treat advanced HER2-positive and AR- positive extramammary Paget disease of the scrotum. It will also learn about the safety of this combination. All patients received Disitamab Vedotin every 2 weeks and Bicalutamide everyday. Follow-up was conducted until disease progression, intolerable adverse reactions occur withdrawal of informed consent by the subject, loss to follow-up, or death. Clinical tumor imaging assessments were performed using RECIST during the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form and comply with the requirements of the protocol.
* Age ≥ 18 years old.
* Confirmed diagnosis by histological examination and/or cytological examination, combined with imaging or ultrasound assessment for mammary and extramammary Paget's disease; pathologically confirmed as HER2 positive, i.e., immunohistochemical test HER2 ≥ 1+, and AR positive, i.e., immunohistochemical test AR ≥ 1+.
* ECOG score: 0 to 1.
* At least one measurable lesion (according to the RECIST criteria, non-nodal lesions with a longest diameter on CT scan ≥10 mm, and nodal lesions with a shortest diameter on CT scan ≥15 mm); or skin lesions that can be evaluated according to the WHO criteria.
* Adequate organ function: Blood routine: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L, Platelet (PLT) ≥70×10^9/L, Hemoglobin (HGB) ≥80g/L; Liver function: Total Bilirubin (TBIL) ≤1.5×Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤3×ULN; Serum Albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN; If the subject has received routine liver protection treatment and meets the above standards, and is stable for at least one week after assessment by the researcher, they may be enrolled; Renal function: Serum Creatinine (Cr) ≤1.5×ULN, or Creatinine Clearance ≥50 mL/min (using the standard Cockcroft-Gault formula): Coagulation function: International Normalized Ratio (INR) ≤1.5 / Prothrombin Time (PT) ≤1.5×ULN, Activated Partial Thromboplastin Time (aPTT) ≤1.5×ULN; - If the subject is receiving anticoagulant therapy, as long as PT and INR are within the range specified for the anticoagulant medication, it is acceptable.
* Estimated life expectancy ≥3 months.

Exclusion Criteria:

* Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Have had active autoimmune diseases within 2 years prior to the start of the study treatment that required systemic treatment (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressants), except for replacement therapies (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency); currently receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy.
* The dose is >10mg/day of prednisone or other equivalent hormones, and it is within 2 weeks of the first administration and still in use;
* Have a history of active tuberculosis;
* Have uncontrollable, recurrent drainage of ascites, pericardial effusion, or pleural effusion;
* Have undergone major organ transplantation;
* Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of the study treatment; or have chronic non-healing wounds or fractures;
* Have a history of live attenuated vaccine administration within 14 days prior to the start of the study treatment or plan to receive live attenuated vaccine vaccination during the study period;
* Have had a severe hypersensitivity reaction after the use of monoclonal antibodies; known allergy to the active ingredients or excipients of this study drug;
* Within 4 weeks prior to the start of the study, are participating in or have participated in other clinical studies;
* Have a history of severe allergies;
* Have a risk of bleeding, or coagulation dysfunction, or are currently receiving -thrombolytic therapy;
* Have a history of substance abuse and are unable to quit or have mental disorders;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study, or there are other reasons deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | every 6 weeks,up to 24 weeks
  ORR includes two categories:
  Complete Response (CR): All target lesions in the patient have completely disappeared, and no new lesions have appeared for a certain time.
  Partial Response (PR): The tumor in the patient has reduced in size by at least 30%, and this reduction has been maintained for a certain period.

SECONDARY OUTCOMES:
Progression free survival | through study completion, an average of 2 year
  Progression-Free Survival (PFS) is a clinical endpoint used primarily in oncology to measure the effectiveness of a treatment in delaying the progression of a disease. It is defined as the length of time during which a patient's disease does not get worse after starting a treatment. PFS takes into account the time from the start of treatment until the first occurrence of disease progression, or the patient's death if it occurs before progression.
advance events | through study completion, an average of 2 year
  advance events

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data is protected.